CLINICAL TRIAL: NCT03381937
Title: Impact of the Pre-phonatory Inspiratory Volume on the Speech Quality of Neuromuscular Patients Dependent on Non-invasive Ventilation
Acronym: PREPHONO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-A00705-48
Record Dates: First submitted 2017-09-21; First posted 2017-12-22 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Neuromuscular Diseases; Non Invasive Ventilation
Keywords: mechanical ventilation; noninvasive ventilation; neuromuscular disorder; phonation; mouthpiece ventilation
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Intervention Model Description: monocentric, open, randomize, crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Spontaneous breathing (No Intervention): Spontaneous breathing without mechanical ventilation
- Conventional mechanical ventilation (Experimental): Conventional mechanical ventilation, with patient ventilator usual parameters
  Interventions: Other: speech trial
- Speech specific mechanical ventilation (Experimental): Mechanical ventilation with specific parameters to improve speech
  Interventions: Other: speech trial

INTERVENTIONS:
Other: speech trial — speech trial during different ventilation conditions
  Arms: Conventional mechanical ventilation; Speech specific mechanical ventilation

SUMMARY:
We want to demonstrate that modifications of the ventilation parameters are liable to improve the different characteristics of phonation (duration, intensity, prosody..) in neuromuscular patients who are dependent on non invasive ventilation.

DETAILED DESCRIPTION:
Speech and communication quality depend on respiration efficiency. The respiratory involvement observed in neuromuscular disorders can impair speech quality in patients, while the underlying disease may also contribute to alter phonation.

Nowadays, the first line treatment of neuromuscular chronic neuromuscular respiratory failure is noninvasive ventilation (NIV). With disease progression, it is used with increasingly duration during daytime. In that situation, mouthpiece ventilation is preferred as it allows efficient ventilation while being more comfortable for patients who can chose when they want to be ventilated. However, in that situation, patients do not receive ventilatory support while they are speaking which puts them in a less favorable situation for speech. We think that pre-phonation inspiratory volume is an essential part of speech quality. Without mechanical ventilation, this volume is reduced as a consequence of respiratory failure but it is liable to increase significantly if the patient used the volume delivered by the ventilator .

We believe that phonation is improved by NIV by applying specific ventilation parameters in patients dependant on mechanical ventilation. The modification could be used by neuromuscular patients to improve speech quality; the patients would then be able to use their usual ventilatory support to improve phonation and modulation of their speech.

In this crossover open labelled, randomised study, done in a single center (home ventilation unit of the referral center of Hospital Raymond Poincaré HUPIFO (University Hospital of Western Paris and Ile de France) (Garches, France)), phonation characteristics will be studied in 3 situations (during spontaneous breathing without ventilatory support, with the usual NIV parameters, with speech-specific NIV parameters) during which speech trials will be performed.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (age > or equal to 18)
* chronic restrictive respiratory failure due to neuromuscular disease
* spontaneous breathing autonomy of at least one hour during the days
* stable clinical state
* patient with middle school education level (able to read)
* patients using life support ventilator ((Astral 150 (ResMed®), Elysée (ResMed®), Trilogy (Philips Respironics®), VentilogicLS (Weinman®), Vivo 40 (Breas®), PB560 ou Légendair (Covidien®), Monal T50 (Air liquide system®))

Exclusion Criteria:

* refusal to participate
* unability to cooperate
* illiterate patients
* tracheostomised patients
* spontaneous breathing autonomy < 1h
* cardiovascular instability
* not registered with the social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-02-06 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Phonation duration | 1 hour
  evaluation by the measurement of the longest duration of a sustained A sound. The subject is asked to sustain a vowel as long as possible during a respiratory cycle while being recorded. Phonation duration is measured (in seconds) on the recording

SECONDARY OUTCOMES:
Speech Intelligibility | 1 hour
  assessment of intelligibility during reading of preselected words by listeners blinded to ventilation condition with a validated scale
Quality of prosodia | 1 hour
  evaluation of prosodia by listeners blinded to ventilation condition with a score based on the number of correct identification
Phonation flow | 1 hour
  Measurement of the number of syllables/min during the reading of a predetermined text
Reading duration | 1 hour
  Measurement of the duration for the reading of a predetermined text
Phonation quality | 1 hour
  evaluation of the phonation quality by the patient with a horizontal visual analogical scale ranked from 0 to 10 (0= very poor quality and 10= very good quality). The scale is 10 cm long ; the patient indicate his perceived sensation on the scale and the according measure (between 0 and 10) is recorded
Breathing quality | 1 hour
  evaluation of the breating quality during speech in each condition by the patient with a horizontal visual analogical scale ranked from 0 to 10 (0= very uncomfortable and 10= very comfortable). The scale is 10 cm long ; the patient indicate his perceived sensation and the according measure (between 0 and 10) is recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Raymond Poincaré hospital, Garches, France

IPD SHARING:
Plan to Share IPD: No